CLINICAL TRIAL: NCT05203887
Title: Short- and Long-term Outcomes of Stenting for Symptomatic Intracranial Arterial Stenosis: a Cohort Study
Status: Completed | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mostafa Abdelmomen Sayed, Assistant lecturer, Sohag University
Other Study IDs: Soh-Med-22-01-10
Record Dates: First submitted 2022-01-13; First posted 2022-01-24 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Atherosclerosis
MeSH Terms: conditions — Intracranial Arteriosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to assess short and long term outcomes of stenting for symptomatic intracranial arterial stenosis.

ELIGIBILITY:
Inclusion Criteria:

* Participants had a symptomatic intracranial stenosis of 70-99 percentage (%) with a lesion length of ≤15 mm and target vessel diameter of ≥2.0 mm in the intracranial internal carotid, middle cerebral, intracranial vertebral or basilar arteries and the measurements of stenosis will be made on magnetic resonance angiography (MRA) using the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) trial method and confirmed by digital subtraction angiography (DSA).
* Presented with transient ischemic attack (TIA) or stroke within the past 12 months attributed to the stenosis.

Exclusion Criteria:

* Participants with acute infarctions within the past 3 weeks.
* Severe arterial tortuosity prevents the deployment of endovascular devices.
* Non-atherosclerotic lesion on magnetic resonance imaging (MRI), embolic or perforator stroke on MRI or computerized tomography (CT).
* A baseline modified Rankin Scale (mRS) score of >3.
* Massive cerebral infarction (>1/2 middle cerebral artery (MCA) territory), intracranial hemorrhage, epidural or sub-dural hemorrhage, and intracranial brain tumor on CT or MRI scan.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic intracranial arterial stenosis caused by intracranial atherosclerosis
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
Cerebrovascular events | 30 days after stenting
  Any stroke (including ischemic or hemorrhagic stroke) or TIA after stenting within the territory of the target vessel.
Death | 30 days after stenting
  Death after stenting within the territory of target vessel.
Cerebrovascular events | 30 days to1 year after stenting
  Ischemic or hemorrhagic stroke within the territory of the target vessel.
Death | 30 days to1 year after stenting
  Vascular death after stenting within the territory of target vessel

SECONDARY OUTCOMES:
Complications | Peri-operative period
  During the peri-operative period, complications such as vasospasms, acute thrombosis, vascular rupture, cerebral infarction, and cerebral haemorrhage will be recorded.
Number of participants with restenosis | 1 year after stenting
  Magnetic resonance angiography (MRA) will be used to calculate the number and incidence of restenosis among all participants.
The degree of restenosis of the target vessel | 1 year after stenting
  The degree of restenosis will be assessed by performing magnetic resonance angiography (MRA) using the Warfarin-Aspirin Symptomatic Intracranial Disease (WASID) trial method for the measurements of arterial stenosis.
Change from baseline in The National Institutes of Health Stroke Scale (NIHSS) score | Baseline and 30 days after stenting
  The National Institutes of Health Stroke Scale (NIHSS) score is a tool used to objectively quantify the impairment caused by a stroke and to evaluate stroke severity. It ranges from 0 to 42, with 42 being the highest and 0 being the lowest. The higher the NIHSS score, the worse the neurological function.
Change from baseline in modified Rankin Scale (mRS) score | Baseline and 30 days after stenting
  The modified Rankin Scale (mRS) score is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.it ranges from 0 to 6 .The higher the mRS score, the worse the prognosis.
Change from baseline in The National Institutes of Health Stroke Scale (NIHSS) score | Baseline and 1 year after stenting
  The National Institutes of Health Stroke Scale (NIHSS) score is a tool used to objectively quantify the impairment caused by a stroke and to evaluate stroke severity. It ranges from 0 to 42, with 42 being the highest and 0 being the lowest. The higher the NIHSS score, the worse the neurological function.
Change from baseline in modified Rankin Scale (mRS) score | Baseline and 1 year after stenting
  The modified Rankin Scale (mRS) score is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke.it ranges from 0 to 6 .The higher the mRS score, the worse the prognosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams university, Cairo, Egypt